CLINICAL TRIAL: NCT05593692
Title: Gender Differences and Age Related Differences in Emergency Department Admission
Acronym: SADE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5121
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Emergencies; Gender; Age Problem
Keywords: sex; gender; age; emergency department
MeSH Terms: conditions — Emergencies; Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about difference related to age and gender in patients admitted to emergency department.

DETAILED DESCRIPTION:
Objectives: Medicine is progressively becoming aware of the clinical difference among patients who present different age, gender, and comorbidities. Our goal is to examine how often different groups of patients access the Emergency Department and for which causes, as well as their different hospitalization and death rates.

Materials and methods: The investigators will collect and analyze data from all patients evaluated at the emergency department of "Fondazione Policlinico Agostino Gemelli" and "Istituto Clinico Humanitas di Milano" from January 2014 to December 2023, the sample obtained will be divided into four groups: younger than 50 years old, 50-65 years old, 66.75 years old, older than 75; each of these groups is divided between males, females and people who do not identify with either of those genders

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 y
* Admitted to emergency department

Exclusion Criteria:

* Age under 18 y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ED
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days
  Death

SECONDARY OUTCOMES:
length of stay | 180 days
  length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Fondazione Policlinico Agostino Gemelli, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No